CLINICAL TRIAL: NCT05910255
Title: An In Depth Study Exploring Patient Experiences of Individuals Participating in Hypertension Clinical Trials
Brief Title: A Detailed Look At What Patients Experience When They Take Part In Hypertension Clinical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 87814554
Record Dates: First submitted 2023-06-09; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research study aims to identify the obstacles faced by specific demographic groups of hypertension patients during their engagement in clinical trials. The study will collect in-depth information from participants and identify common factors that impede their enrollment or successful completion of these trials.

By examining data from various demographic perspectives, the study aims to identify patterns impacting future hypertension patients' experiences.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Diagnosis of hypertension
* Ability to understand the study procedures, benefits and risks, and sign a written informed consent document.

Exclusion Criteria:

* Enrolled in another research study
* Inability to provide written informed consent
* Women of childbearing potential without a negative pregnancy test; or women who are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertension who are actively participating in a clinical research, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of hypertension patients who decide to join in a clinical study | 3 months
Rate of patients who remain in a hypertension clinical study to completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Margolis KL, Crain AL, Green BB, O'Connor PJ, Solberg LI, Beran M, Bergdall AR, Pawloski PA, Ziegenfuss JY, JaKa MM, Appana D, Sharma R, Kodet AJ, Trower NK, Rehrauer DJ, McKinney Z, Norton CK, Haugen P, Anderson JP, Crabtree BF, Norman SK, Sperl-Hillen JM. Comparison of explanatory and pragmatic design choices in a cluster-randomized hypertension trial: effects on enrollment, participant characteristics, and adherence. Trials. 2022 Aug 17;23(1):673. doi: 10.1186/s13063-022-06611-3. PMID 35978336
- [Background] Noone C, Dwyer CP, Murphy J, Newell J, Molloy GJ. Comparative effectiveness of physical activity interventions and anti-hypertensive pharmacological interventions in reducing blood pressure in people with hypertension: protocol for a systematic review and network meta-analysis. Syst Rev. 2018 Aug 21;7(1):128. doi: 10.1186/s13643-018-0791-9. PMID 30131071
- [Background] Cimmaruta D, Lombardi N, Borghi C, Rosano G, Rossi F, Mugelli A. Polypill, hypertension and medication adherence: The solution strategy? Int J Cardiol. 2018 Feb 1;252:181-186. doi: 10.1016/j.ijcard.2017.11.075. Epub 2017 Nov 23. PMID 29180263

DOCUMENTS (1):
  • Informed Consent Form (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT05910255/ICF_000.pdf